CLINICAL TRIAL: NCT01948622
Title: Anxiety Control by Using Erythrina Mulungu in Mandibular Third Molars Extraction
Brief Title: Anxiety Control by Erythrina Mulungu
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Liane Maciel de Almeida Souza (Other)
Collaborators: University of Campinas, Brazil (Other)
Responsible Party: Sponsor-Investigator, Liane Maciel de Almeida Souza, Assistant Professor, Universidade Federal de Sergipe
Organization: Universidade Federal de Sergipe (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mulungu-401-2011
Record Dates: First submitted 2013-09-10; First posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Dental Anxiety; Impacted Third Molar Tooth
Keywords: Anxiety; Third molar surgery; Blood pressure; Heart rate; Oxygen saturation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mulungu (Active Comparator): 500 mg Mulungu Matusa® (Erytrina mulungu, 2 capsules of 250 mg) administered v.o., one hour before the surgical procedure.
  Interventions: Drug: Mulungu
- placebo (Placebo Comparator): 500 mg of starch (2 capsules of 250 mg) administered v.o., one hour before the surgical procedure.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mulungu — 500 mg/single dose/1 hour before dental surgery
  Other Names: Mulungu Matusa, Erytrina mulungu
  Arms: Mulungu
Drug: Placebo — 500 mg/single dose/1 hour before dental surgery
  Arms: placebo

SUMMARY:
This study evaluated the effectiveness of the Erythrina mulungu in controlling anxiety in patients undergoing bilateral extraction of asymptomatic, impacted mandibular third molars.

DETAILED DESCRIPTION:
: In this research, characterized as a randomized, double-blind, crossover study, 30 healthy volunteered patients (05 men and 25 women) aged 18 or older who received a capsule of 500mg of Mulungu Matusa ® or placebo, orally, one hour before the procedure were selected. The level of anxiety was assessed through questionnaires and physical parameters, such as blood pressure, heart rate and oxygen concentration. Data were collected, tabulated and analyzed by the following statistical tests: chi-square, t-test, ANOVA and Tukey test, Friedman, Fisher's exact test with significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* indication of bilateral extraction of asymptomatic, impacted mandibular third molars

Exclusion Criteria:

* patients under the age of 18
* any general health problem based on the medical history and physical examination
* history of use of any medication within 15 days before the beginning of the research
* history of hypersensitivity to drugs, substances or materials used in this experiment
* pregnancy or lactation
* history of pericoronitis

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Changes in anxiety report | Change from baseline to 7 days
  Changes in the subjects' anxiety level was observed by using a Modified Corah Dental Anxiety Scale in three times: at baseline, in the day of surgery and after 7 days of the procedure.

SECONDARY OUTCOMES:
Changes in blood pressure | Change from baseline to 2 hours
  blood pressure (mmHg) was measured before drug administration, 30 minutes after drug administration and during local anesthesia, incision, tooth removal and suturing.
Changes in heart rate | Change from baseline to 2 hours
  heart rate (bpm) was measured before drug administration, 30 minutes after drug administration and during local anesthesia, incision, tooth removal and suturing.
Changes in oxygen saturation | Change from baseline to 2 hours
  oxygen saturation (SpO2) was measured before drug administration, 30 minutes after drug administration and during local anesthesia, incision, tooth removal and suturing.

CONTACTS AND LOCATIONS:
Overall Officials: Liane M Souza, PhD, Principal Investigator — Federal University of Sergipe
Locations (1):
- Federal University of Sergipe, Aracaju, Sergipe, Brazil

REFERENCES:
- [Background] Balbani AP, Silva DH, Montovani JC. Patents of drugs extracted from Brazilian medicinal plants. Expert Opin Ther Pat. 2009 Apr;19(4):461-73. doi: 10.1517/13543770902824180. PMID 19441926
- [Background] Flausino OA Jr, Pereira AM, da Silva Bolzani V, Nunes-de-Souza RL. Effects of erythrinian alkaloids isolated from Erythrina mulungu (Papilionaceae) in mice submitted to animal models of anxiety. Biol Pharm Bull. 2007 Feb;30(2):375-8. doi: 10.1248/bpb.30.375. PMID 17268084
- [Background] Flausino O Jr, Santos Lde A, Verli H, Pereira AM, Bolzani Vda S, Nunes-de-Souza RL. Anxiolytic effects of erythrinian alkaloids from Erythrina mulungu. J Nat Prod. 2007 Jan;70(1):48-53. doi: 10.1021/np060254j. PMID 17253849
- [Background] Onusic GM, Nogueira RL, Pereira AM, Flausino Junior OA, Viana Mde B. Effects of chronic treatment with a water-alcohol extract from Erythrina mulungu on anxiety-related responses in rats. Biol Pharm Bull. 2003 Nov;26(11):1538-42. doi: 10.1248/bpb.26.1538. PMID 14600397